CLINICAL TRIAL: NCT04670666
Title: National, Multicenter, Randomized, Double-blind, Triple-dummy, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Madalena Association in the Treatment of Type II Diabetes Mellitus.
Brief Title: Efficacy and Safety of Madalena Association in the Treatment of Type II Diabetes Mellitus
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS1419 - MADALENA
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; empagliflozin; Linagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MADALENA (Experimental): The study is triple-dummy. The patient must take 3 tablets once a day, as follows:
  1 tablet Madalena association, oral;
  1 tablet empagliflozin + linagliptin association placebo, oral;
  1 tablet metformin placebo, oral.
  Interventions: Drug: MADALENA ASSOCIATION; Other: METFORMIN PLACEBO; Other: EMPAGLIFLOZIN + LINAGLIPTIN PLACEBO
- Metformin + empagliflozin + linagliptin (Active Comparator): The patient must take 3 tablets once a day, as follows:
  1 tablet Madalena association placebo, oral;
  1 tablet empagliflozin + linagliptin association, oral;
  1 tablet metformin, oral.
  Interventions: Drug: METFORMIN; Drug: EMPAGLIFLOZIN + LINAGLIPTIN; Other: MADALENA ASSOCIATION PLACEBO

INTERVENTIONS:
Drug: MADALENA ASSOCIATION — Madalena association coated tablet.
  Arms: MADALENA
Drug: METFORMIN — Metformin 1000 mg extended-release tablet.
  Arms: Metformin + empagliflozin + linagliptin
Drug: EMPAGLIFLOZIN + LINAGLIPTIN — Empagliflozin 10 mg + linagliptin 5 mg coated tablet.
  Arms: Metformin + empagliflozin + linagliptin
Other: MADALENA ASSOCIATION PLACEBO — Madalena association placebo tablet.
  Arms: Metformin + empagliflozin + linagliptin
Other: METFORMIN PLACEBO — Metformin placebo tablet.
  Arms: MADALENA
Other: EMPAGLIFLOZIN + LINAGLIPTIN PLACEBO — Empagliflozin + linagliptin placebo tablet.
  Arms: MADALENA

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Madalena association in the treatment of type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the informed consent forms;
* Participants with 18 years of age or greater;
* Participants presenting the diagnosis of type II diabetes mellitus, and who did not reach the therapeutic goals of HbA1c with previous dietary, physical exercise guidance and at least 3 months with two anti-hyperglycemic agents (dual therapy);
* HbA1c ≥ 7,5% and ≤ 10,5% and fasting blood glucose > 100 mg/dL at the screening visit;
* BMI (body mass index) > 19 Kg/m2 and ≤ 45 Kg/m2.

Exclusion Criteria:

* Any clinical and laboratory findings that, in the judgment of the investigator, may interfere with the safety of research participants;
* History of alcohol abuse or illicit drug use;
* Participation in a clinical trial in the year prior to this study;
* Pregnancy or risk of pregnancy and lactating patients;
* Known hypersensitivity to the formula components used during the clinical trial;
* Type 1 diabetes mellitus;
* Fasting blood glucose > 300 mg/dL;
* Risk factors for volume depletion;
* Impaired renal function and end-stage renal disease;
* Participants with current treatment and continued for more than 15 days with systemic steroids at the time of informed consent;
* Impaired hepatic function;
* Medical history of pancreatic diseases that may suggest insulin deficiency;
* Bariatric surgery in the last two years and/ or other gastrointestinal surgeries that can cause chronic malabsorption syndrome;
* Condition that, in the investigator's judgment, may favor clinically significant changes in CPK levels;
* Medical history of acute coronary syndrome, stroke, unstable congestive heart failure, or respiratory failure within 6 months prior to informed consent;
* Current medical history of cancer and/ or cancer treatment in the last 5 years;
* Medical history of metabolic acidosis and/or using drugs that may cause lactic acidosis;
* Medical history of blood dyscrasia or any other hemolytic disorders;
* Participants using sulfonylureas and/or insulin therapy;
* Treatment with anti-obesity drugs for less than 2 months or with dose change in the last 2 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in glycated hemoglobin (HbA1c) levels. | 120 days

SECONDARY OUTCOMES:
Incidence and severity of adverse events recorded during the study. | 150 days

CONTACTS AND LOCATIONS:
Locations (1):
- EMS, Hortolândia, São Paulo, Brazil